CLINICAL TRIAL: NCT00066898
Title: "Reduction of Vascular Inflammation and Coronary Atherosclerosis With AGI-1067, a V-Protectant, Reduces Cardiovascular Events in Patients With Coronary Artery Disease"
Brief Title: ARISE - Aggressive Reduction of Inflammation Stops Events
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AtheroGenics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AGI-1067/042
Record Dates: First submitted 2003-08-06; First posted 2003-08-08 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-09

CONDITIONS: Atherosclerosis; Coronary Artery Disease; Myocardial Infarction; Unstable Angina
Keywords: succinobucol; AGI-1067; coronary artery disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Myocardial Infarction; Angina, Unstable | interventions — succinobucol

INTERVENTIONS:
Drug: AGI-1067

SUMMARY:
To assess the safety and efficacy of AGI-1067, as compared to placebo, in the treatment of vascular inflammation and atherosclerosis by assessing the reduction in cardiovascular events.

DETAILED DESCRIPTION:
This study will be a Phase III multi-center, double-blind, parallel group, placebo-controlled trial involving approximately 260 study sites in the United States, Canada, South Africa and the United Kingdom. It is expected that approximately 6,600 subjects will be screened in order to randomize approximately 6,000 subjects globally (3,000 in each arm of the study). Male or female subjects with coronary artery disease are eligible to participate if they meet all required inclusion and exclusion criteria. Recruitment will be delayed for one month in subjects who have had a PCI. Subjects who have a PCI planned at the time of screening or randomization, will not be randomized until one month after this planned PCI has been conducted. All subjects who successfully complete the screening phase and meet all required inclusion and exclusion criteria will be entered into the single-blind, placebo Run-In phase of the study to establish compliance. The placebo Run-In medication will be identical to the blinded study drug used in the randomized portion of the study. After the completion of the two-week Run-In, if compliance has been adequate, study subjects will be randomized to receive AGI-1067 300 mg (two 150 mg tablets daily with a meal) or placebo (approximately equal numbers of subjects per treatment group) for a minimum of 12 months. It is anticipated that subject accrual will occur over a period of approximately 24 months and that all subjects will be followed until at least 990 subjects have experienced a primary event. Subjects will remain on drug therapy from randomization until the end of the study. It is estimated that the first subject recruited will be exposed to blinded therapy for 30 to 36 months, and the last subject will be exposed for a minimum of 6 to 12 months. For the purposes of this study one month will be equal to 28 days. The subject will be asked to return to the clinic at 1 month, 3 months, and every 3 months thereafter during the treatment phase. All clinical laboratory procedures and electrocardiographic interpretations will be performed by central laboratories. Over the study period, subjects will be followed for the occurrence of major adverse cardiovascular events. These potential endpoints will be adjudicated by an independent endpoint committee. This committee will consist of cardiologists and other physician reviewers who will be blinded to the treatment. For the purposes of safety, the trial will be monitored by an independent Data Safety Monitoring Board. This Board will consist of Cardiologists, and at least one Statistician experienced in the conduct of clinical trials. The Board will meet approximately every 6 months to review subject safety data.

ELIGIBILITY:
IRB-approved informed written consent must be provided by all subjects prior to screening and study entry.

A. Inclusion Criteria

1. Informed written consent from the subject prior to Screening
2. Acute MI or unstable angina not less than 14 days and not more than one year prior to randomization
3. Male or female subjects in one of the two following groups:

   1. Subjects with diabetes mellitus (NIDDM or IDDM) 18 years of age or older
   2. Subjects (without diabetes mellitus) 55 years of age or older with one of the following additional risk factors:

   (i) Age 60 or older (ii) Low HDL-C as evidenced by: Male: HDL-C < 40 mg/dL or Female: HDL-C < 50 mg/dL (iii) Previous Myocardial Infarction (in addition to the index event), or diagnosis of Atherosclerosis in a non-coronary vessel (e.g. history of prior stroke, presence of PVD) (iv) Prior history of CHF (Congestive Heart Failure) or ejection fraction < 40%
4. Females must be non-lactating and not of child bearing potential

B. Exclusion Criteria

1. Subjects who are hemodynamically or clinically unstable
2. Subjects who have had a PCI in the last 30 days
3. Subjects who have had coronary artery bypass (CABG) in the last 3 months
4. Subjects on a waiting list for revascularization or revascularization already planned
5. Current symptoms consistent with moderate or severe CHF despite medical therapy
6. Clinically significant valvular heart disease or Hypertrophic Obstructive Cardiomyopathy
7. Uncontrolled hypertension (e.g., sitting systolic BP > 180 mm Hg on antihypertensive therapy)
8. Known major hematologic, renal, hepatic, metabolic, gastrointestinal or endocrine dysfunction
9. Subjects taking and requiring continued therapy with drugs known to significantly prolong the QT interval (this will not include drugs associated with minor effect on the QT interval of less than 15 msec.)
10. Life-threatening illness where the subject is not expected to survive for 2 years or any history of cancer or malignancy within the past 5 years except for basal cell carcinoma or squamous cell carcinoma of the skin
11. A history of intolerance to probucol (Lorelco™)
12. Unreliability as a study participant based on the Investigator's (or designee's) knowledge of the subject (e.g., alcohol or other drug abuse, inability or unwillingness to adhere to the protocol, or psychosis)
13. Participation in any investigational drug study within 30 days prior to study entry, or expectation to participate in any other investigational drug study during the course of the ARISE study.
14. Previous participation in a study involving AGI-1067

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000
Dates: Start 2003-06; Study Completion 2006-12

PRIMARY OUTCOMES:
Length of time to the first occurrence of one of six adjudicated events: cardiovascular mortality, resuscitated cardiac arrest, non-fatal MI, non-fatal stroke, hospitalization for angina pectoris, or use of coronary revascularization.

SECONDARY OUTCOMES:
Time to first incidence of any of the following: all cause mortality, resuscitated cardiac arrest, non-fatal MI, non-fatal stroke, use of coronary revascularization, and hospitalization for unstable angina
Time to first incidence of any of the following: cardiovascular mortality, resuscitated cardiac arrest, non-fatal MI, non-fatal stroke, and hospitalization for unstable angina
Time to first incidence of any of the following: cardiovascular mortality, resuscitated cardiac arrest, non-fatal MI, and non-fatal stroke

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Pfeffer, MD, Study Chair — Cardiovascular Division Brigham and Women's Hospital; Jean-Claude Tardif, MD, Study Chair — Montreal Heart Institute; John McMurray, MD, Principal Investigator — Western Infirmary; Eric Klug, MD, Principal Investigator — Independent Medical Practitioner - South Africa
Locations (219):
- United States (128):
  - Cardiovascular Associates, Birmingham, Alabama
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - The Heart Center/Oracle Research, Huntsville, Alabama
  - Tri City Cardiology Consultants, Mesa, Arizona
  - Tri-City Cardiology Consultants, Mesa, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Lovelace Scientific Resources, Phoenix, Arizona
  - Sonoran Health Specialists, Scottsdale, Arizona
  - Capitol Interventional Cardiology, Carmichael, California
  - Escondido Cardiology, Escondido, California
  - Merced Heart Associates, Merced, California
  - Orange County Research Cntr, Orange, California
  - ARI Clinical Trials, Redondo Beach, California
  - Radiant Research, Santa Rosa, California
  - Pikes Peak Cardiology, Colorado Springs, Colorado
  - Aurora Denver Cardiololgy Associates, Denver, Colorado
  - Heart and Vascular Clinic N CO, Fort Collins, Colorado
  - Connecticut Clinical Research, Bridgeport, Connecticut
  - Cardiac Specialists, PC, Trumbull, Connecticut
  - Christiana Care Health Svcs, Newark, Delaware
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - SW Florida Heart Group, Fort Myers, Florida
  - Univ of Florida, Cardiology, Gainesville, Florida
  - Diagnostic Cardiology, Jacksonville, Florida
  - Jacksonville Cntr Clin Research, Jacksonville, Florida
  - Jacksonville Heart Center, Jacksonville Beach, Florida
  - Watson Clinic LLP, Lakeland, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Orlando Heart Cntr, Orlando, Florida
  - Cardiovascular Cntr of Sarasota, Sarasota, Florida
  - The Broward Heart Group, Tamarac, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Crawford Long Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Fuqua Hrt Cntr Piedmont Hosp, Atlanta, Georgia
  - Harbin Clinic, Rome, Georgia
  - Idaho Cardiology Associates, Boise, Idaho
  - Heart Care Research Foundation, Blue Island, Illinois
  - Peryam and Kroll Healthcare, Chicago, Illinois
  - Heartcare Midwest Heart Inst, Peoria, Illinois
  - The Heart Group, Evansville, Indiana
  - Welborn Clinic Research Center, Evansville, Indiana
  - Parkview Hospital, Fort Wayne, Indiana
  - Care Group St. Vincent Hosp of IN, Indianapolis, Indiana
  - Research Inst of Middle America, Jeffersonville, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - Univ of IA College of Medicine, Iowa City, Iowa
  - Research Inst of Kansas Inc, Wichita, Kansas
  - Cardiovascular Associates, Louisville, Kentucky
  - Louisiana Heart Center, Chalmette, Louisiana
  - The Office of Dr. Richard Gilmore, Lake Charles, Louisiana
  - Heart Clinic of Louisiana, Marrero, Louisiana
  - Cardiovascular Inst of the South, Morgan City, Louisiana
  - Cardiovascular Inst of the South, New Iberia, Louisiana
  - Louisiana Clinical Trials, New Orleans, Louisiana
  - Tulane Univ Medical Center, New Orleans, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Cardiovascular Inst of South, Thibodaux, Louisiana
  - Androscoggin Cardiology, Auburn, Maine
  - Midatlantic Cardiovascular Associates, Baltimore, Maryland
  - Midatlantic Cardiovascular, Baltimore, Maryland
  - Midatlantic Cardiovascular, Bel Air, Maryland
  - Patuxent Medical Group, Columbia, Maryland
  - MD Med Research Ong Med Cntr, Oxon Hill, Maryland
  - Midatlantic Cardiovascular, Towson, Maryland
  - Midatlantic Cardiovascular, Westminster, Maryland
  - Compass Medical Associates, Abington, Massachusetts
  - Gary Brockington, MD, Boston, Massachusetts
  - Lahey Clinic Med Cntr, Burlington, Massachusetts
  - Pentucket Med Assoc Inc, Haverhill, Massachusetts
  - Charles River Med Associates, Natick, Massachusetts
  - Professional Clinical Research, Cadillac, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - The Office of Dr. Keith Pierce, Livonia, Michigan
  - Beaumont Medical Office Bldg, Royal Oak, Michigan
  - Michigan Heart Group, Troy, Michigan
  - St Paul Heart Clinic, Saint Paul, Minnesota
  - N'Touch Research, Kansas City, Missouri
  - St Louis Univ Div Solutions, St Louis, Missouri
  - St Louis Univ Hospital, St Louis, Missouri
  - Washington Univ School of Med, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Creighton Cardiac Center, Omaha, Nebraska
  - Nebraska Heart Institute, Papillion, Nebraska
  - Cardiovascular Assoc of Delaware Valley, Elmer, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - SUNY Downstate Health Science Ctr, Brooklyn, New York
  - St Vincent's Med Cntr NY, New York, New York
  - SUNY Upstate Medical Univ, Syracuse, New York
  - Syracuse Preventive Cardiology, Syracuse, New York
  - Buffalo Cardiology and Pulmonary Associates, Williamsville, New York
  - Mid Carolina Cardiology Research Div, Charlotte, North Carolina
  - City Cardiology Associates, Akron, Ohio
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Sterling Research Group, Cincinnati, Ohio
  - North Ohio Heart Center, Sandusky, Ohio
  - Bluestem Cardiology, Bartlesville, Oklahoma
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Consultants, Tulsa, Oklahoma
  - The Heart Care Group, Allentown, Pennsylvania
  - Tri-State Medical Group, Beaver, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Kandra, Fierer, Kuskin Associates, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Banksville Medical, Pittsburgh, Pennsylvania
  - Rhode Island Cardiovascular Group, Woonsocket, Rhode Island
  - Charleston Cardiology, Charleston, South Carolina
  - Internal Medicine of Greer, Greer, South Carolina
  - Alpha Clinical Research, Clarksville, Tennessee
  - Cardiovascular Research Foundation, Knoxville, Tennessee
  - Amarillo Heart Clinical Research Institute, Amarillo, Texas
  - Pharma Tex Research, Amarillo, Texas
  - Austin Heart PA, Austin, Texas
  - Southeast Texas Cardiology Associates II, Beaumont, Texas
  - Clinical Cardiovascular Research Cntr, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - Research Clinic, Nassau Bay, Texas
  - Sioco Cardiology, PA, San Antonio, Texas
  - Heart Center, Salt Lake City, Utah
  - IHC Health Services, Salt Lake City, Utah
  - DUCCS Research of S Boston, South Boston, Virginia
  - Daniel Gottlieb MD PS, Burien, Washington
  - U of WA NW Lipid Research Cntr, Seattle, Washington
  - Appleton Heart Inst, Appleton, Wisconsin
  - Wisconsin Center for Clinical Research, Elkhorn, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Canada (54):
  - Foothills Hospital Cardiology Div, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - West Coast Cardiology Research, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - St Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre Div of Cardiology, St. John's, Newfoundland and Labrador
  - Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia
  - Halton Heart Institute, Burlington, Ontario
  - The Office of Dr. Syan Gurcharan, Greater Sudbury, Ontario
  - St Joseph Health Care Hamilton, Hamilton, Ontario
  - Kingston Heart Clinic, Kingston, Ontario
  - London Health Sci Cntr Site, London, Ontario
  - Mount St. Joseph's, London, Ontario
  - Newmarket Cardiology Research, Newmarket, Ontario
  - Heart Care Research, Oshawa, Ontario
  - Ottawa Cardiovascular Center, Ottawa, Ontario
  - Vexler Health Services, Ottawa, Ontario
  - Cliks Medical Research, Thunder Bay, Ontario
  - Thunder Bay Regional Health Science Ctr, Thunder Bay, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook and Women's College, Toronto, Ontario
  - University Health Network - Toronto Western Hosp, Toronto, Ontario
  - CMGC-GRID Complexe Hosp, Chicoutimi, Quebec
  - Q & T Research Outaouais, Gatineau, Quebec
  - Recherches Cliniques Theradev, Granby, Quebec
  - The Office of Dr. Jean-Robert Timothee, Greenfield Park, Quebec
  - ViaCar Recherche Clinique, Greenfield Park, Quebec
  - Hosp Regional de Lanaudiere, Joliette, Quebec
  - Cite de la Sante de Laval, Laval, Quebec
  - Clinique de Cardiologie de Levis, Lévis, Quebec
  - Medicayeb, Inc., Longueuil, Quebec
  - ViaCar Recherche Clinique Inc., Longueuil, Quebec
  - CHUM Hopital Notre Dame, Montreal, Quebec
  - CUSM Montreal General Hosp, Montreal, Quebec
  - Hopital du Sacre Coeur De Montreal, Montreal, Quebec
  - Maisonneuve Rosemont Hosp, Montreal, Quebec
  - McGill Univ Health Cntr, Montreal, Quebec
  - Medi-Recherche Inc., Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Recherches Clinicar, Québec, Quebec
  - Cntr Hospital Beauce Etchemin, Saint George, Quebec
  - Reseau Sante Richelieu Yamaska, Saint-Hyacinthe, Quebec
  - Hopital du Haut-Richelieu, Saint-Jean-sur-Richelieu, Quebec
  - Zoom International, Saint-Jérôme, Quebec
  - Neufort Inc., Saint-Lambert, Quebec
  - London Clinical Research, Sherbrooke, Quebec
  - Laval Hospital Pavillion 2U, Ste-Foy, Quebec
  - Cntr Hospitalier Pierre Le Gardeur, Terrebonne, Quebec
  - Centre Hospitalier de Val d'Or, Val-d'Or, Quebec
  - Societe des internistes Bois Fran, Victoriaville, Quebec
  - Pasqua Hosp Coronary Care Unit, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Saskatoon Medical Specialists, Saskatoon, Saskatchewan
- South Africa (19):
  - Dr. Johann Viljoen, Bloemfontein, BLM
  - Fichmed 5, Rosepark Hospital, Bloemfontein, BLM
  - Universitas Hospital, Bloemfontein, BLM
  - 228 Panorama Medi Clinic, Panorama, CT
  - Panorama Medical Clinic, Panorama, CT
  - Tygerberg Hospital, Parow, CT
  - Vincent Pallotti Hospital, Pinelands, CT
  - Vergelegen Medical Clinic, Somerset West, CT
  - Chatsmed Garden Hospital, Chatsworth, DBN
  - Chatsmed Hospital, Chatsworth, DBN
  - 403 Maxwell Centre, Durban, DBN
  - United House, Fordsburg, JHB
  - The Boulders Shopping Center, Halfway House, JHB
  - Mulbarton Medical Center, Mulbarton, JHB
  - Olivedale Clinic, Olivedale, JHB
  - Sunninghill Hospital, Sunninghill, JHB
  - Pretoria Heart Hospital, Arcadia, PTA
  - Unitas Hospital, Lyttelton Centurion, PTA
  - Wilgers Medical Consortium, The Willows, PTA
- United Kingdom (18):
  - King's College Hospital NHS Trust, London, England
  - Barking, Havering & Redbridge Hospital NHS Trust, Romford, Essex
  - Grampian University Hospitals NHS Trust, Aberdeen
  - Sandwell & West Birmingham City Hospital NHS Trust, Birmingham
  - Papworth Hospital NHS Trust, Cambridge
  - The Lothian University Hospitals NHS Trust, Edinburgh
  - North Glasglow University Hospitals NHS Trust, Glasglow
  - South Glasglow University Hospital NHS Trust, Glasglow
  - Western Infirmary Glaglow, Glasglow
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Liverpool NHS Trust, Liverpool
  - South Manchester University Hospitals NHS Trust, Manchester
  - Argyll & Clyde NHS Trust, Paisley
  - Sheffield Teaching Hospitals NHS Trust, Sheffield
  - Forth Valley Acute Hospitals NHS Trust, Stirling
  - University Hospitals of North Staffordshire NHS Trust, Stoke-on-Trent
  - Mid Yorkshire Hospitals, Wakefield

REFERENCES:
- [Derived] Tardif JC, McMurray JJ, Klug E, Small R, Schumi J, Choi J, Cooper J, Scott R, Lewis EF, L'Allier PL, Pfeffer MA; Aggressive Reduction of Inflammation Stops Events (ARISE) Trial Investigators. Effects of succinobucol (AGI-1067) after an acute coronary syndrome: a randomised, double-blind, placebo-controlled trial. Lancet. 2008 May 24;371(9626):1761-8. doi: 10.1016/S0140-6736(08)60763-1. PMID 18502300